CLINICAL TRIAL: NCT01252303
Title: The Effect of a Behavioral Weight Loss Program With Nutrisystem Meal Provision on Change in Weight, Fasting Blood Glucose, Cholesterol, and Blood Pressure Over 12 Weeks.
Brief Title: The Effect of Nutrisystem Meal Provision on Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: Nutrisystem, Inc. (Industry)
Responsible Party: Kelly Webber, assistant professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0639-F3R
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Obesity
Keywords: Obesity, weight loss, meal replacements
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrisystem (Experimental): Group will receive Nutrisystem meals in addition to the behavioral weight loss program.
  Interventions: Behavioral: Nutrisystem
- Control (Active Comparator): Group will receive a behavioral weight loss program only.
  Interventions: Behavioral: Nutrisystem

INTERVENTIONS:
Behavioral: Nutrisystem — Nutrisystem meal replacements for 12 weeks
  Other Names: Weight loss trial

SUMMARY:
The study is to determine the effect of a behavioral weight loss program supplemented with Nutrisystem meal replacements on weight, blood pressure, fasting blood glucose, and blood lipids levels over 12 weeks.

DETAILED DESCRIPTION:
Specific Aim 1- Compare two programs, a standard Internet weight loss program and an Internet behavioral weight loss program, enhanced with Nutrisystem meal provision, on their effectiveness in producing weight loss and improvements in fasting blood glucose, blood pressure, and blood lipid levels over 12 weeks.

Specific Aim 2- Determine the usage and acceptability of the two programs.

Overall Hypothesis:

The Internet program with Nutrisystem meal provision will produce greater improvements in participant's health (weight, blood pressure, blood lipids, and fasting blood glucose) than the standard Internet program alone at 12 weeks. The acceptability and usage of each program will directly correlate with weight loss in participants.

Recruitment Methods Participants will be recruited through advertisements in local newspapers. Randomization A two-group randomized design will be used. After meeting all exclusion/inclusion criteria, completion of all study measurements, and provision of written consent, individuals will be randomized to one of the two study groups: (1) the standard Internet behavioral weight loss program alone or (2) the standard Internet program plus Nutrisystem meal provision.

Timeline and Milestones Recruitment advertisements for the study will be placed in mid-December. Participants who meet all inclusion/exclusion criteria will be invited to a study information session the first week of January.

Delivery Phase (Jan.-April 2011) The delivery phase will entail: (1) conducting study information sessions; (2) baseline assessments; (3) conducting the 12-week Intervention; (4) 12-week assessments. Dr. Webber will conduct study information sessions for qualified participants during the first week of January. Interested participants will then be asked to sign consent forms, fill out motivation questionnaires, and to schedule appointments at the Clinical Research Center (CRC) at the University of Kentucky for baseline assessments of height, weight, waist circumference, blood pressure, fasting blood glucose and blood lipids.

Once measurements at the CRC are taken, participants will be randomized to study group. At baseline each group will receive a 2-hour weight loss group session with a registered dietitian. The weight loss session will include presentation of information on exercise and dietary recommendations, an overview of energy balance, and instructions for self-monitoring, good dietary practices, exercise safety recommendations, and orientation to the study website.

Both groups will be given password protected access to a standard Internet program. The website will include 12 weekly lessons based on the Diabetes Prevention Program (DPP), a message board feature, a link to a personal self-monitoring diary, a library of links to diet, exercise, and behavioral resources available on the web, and a weekly weight loss tip. The Nutrisystem group will receive 2 weeks of meals at the baseline 2-hour session. They will be asked to return every two weeks to the clinic to pick up Nutrisystem meals.

Evaluation Phase (May-Oct. 2011) The evaluation phase of the project will entail: (1) data entry, cleaning and analysis; (2) final report preparation; (3) manuscript preparation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must (1) be age 25 to 65 years old; (2) have a BMI of > 30 and <45; (3) own a home computer with access to the Internet.

Exclusion Criteria:

* Participants must not: (1) have a medical diagnosis of orthopedic or joint problems that may prohibit regular exercise; (2) endorse any of the first three items on the Physical Activity Readiness Questionnaire (PAR-Q): heart problems, chest pain, faintness or dizzy spells; (3) endorse any of the other items on the PAR-Q without a physician's consent; (4) have had a hospitalization for a psychiatric disorder within the last year; (5) have a history of anorexia or bulimia nervosa; (6) have a medical diagnosis of cancer or HIV with the exception of skin cancer; (7) have a diagnosis with a major psychiatric disorder (i.e. bipolar disorder or schizophrenia); (8) be pregnant, nursing, or planning to become pregnant within the study period; (9) be less than 9 months post-partum; (10) have a recent weight loss of > 10 pounds; (11) be using centrally-active medications, with the exception of alcohol and caffeine.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
weight change | 12 weeks
  Amount of weight lost in the 12 week study.

SECONDARY OUTCOMES:
Blood pressure | 12 weeks
  The change in blood pressure over the 12 weeks.
Fasting Blood Glucose | 12 weeks
  Change in fasting blood glucose over the 12 weeks.
blood lipids | 12 weeks
  Change in blood lipids over the 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly H Webber, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States